CLINICAL TRIAL: NCT02792556
Title: Evaluation of Urine Pregnancy Test, CHECK TOP Test, Compared to Transvaginal Ultrasound During Control Visit Post Drug Abortion (CHECK-TOP).
Brief Title: Urine Pregnancy Test Compared to Transvaginal Ultrasound (CHECK-TOP).
Acronym: CHECK-TOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0263
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Drug Abortion
Keywords: drug abortion; urine pregnancy test; negative predictive value; check Top test; transvaginal ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patient having a drug abortion: Urine pregnancy test for adult women having a drug abortion until 8 weeks of amenorrhea, presenting to the control visit between the 14th and 21th day after drug intake.
  Interventions: Device: Urine pregnancy test

INTERVENTIONS:
Device: Urine pregnancy test — Urine pregnancy test Check Top after transvaginal ultrasound

SUMMARY:
According to a study of the DREES (Direction de la Recherche, des Etudes, de l'Evaluation et des Statistiques), in 2013, nearly 229 000 abortions were performed in France, an increasing number.

The success rate of drug abortion before 49 days of amenorrhea, defined by the National Health Autority as a complete abortion not requiring surgery, varies from 92 to 98% depending on the pregnancy term and the dose used.

The control visit is performed between the 14th day and the 21th day post abortion. Its role is to monitor the effectiveness of the method, to verify absence of complication and to better adapt contraception to prevent another unwanted pregnancy. The choice of the method is left to the physician's discretion: β-HCG dosage, pelvic or transvaginal ultrasound.

In the Orthogenic Departement of the Croix-Rousse Hospital Lyon, France, the method performed during the control visit is transvaginal ultrasound.

To simplify the monitoring of drug abortion, a urine pregnancy test would be an attractive alternative to transvaginal ultrasound: simplicity of use, speed, ease of interpretation and low cost.

The main objective of this study is to evaluate the diagnostic value of urine pregnancy test CHECK TOP compared to transvaginal ultrasound in monitoring the outcome of drug abortion during the control visit.

This is a monocentric observational study.

ELIGIBILITY:
* Inclusion Criteria:

  * Women ≥18 years of age
  * Undergoing drug abortion in Orthogenic Departement, Croix-Rousse Hospital, Lyon
  * Intrauterine pregnancy, single or multiple, until 8 weeks of amenorrhea
  * Agreeing to participate in the study after receiving information note
  * Affiliated to a social security system
  * Not subject to a measure of legal protection
* Exclusion Criteria:

  * Women <18 years
  * Ineligible patient to drug abortion
  * Patient practicing a surgical abortion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult women having a drug abortion until 8 weeks of amenorrhea, presenting to the control visit between the 14th and 21th day after drug intake.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value of urine pregnancy test CHECK TOP | During control visit post drug abortion, after transvaginal ultrasound (at day14 or day21)
  Negative predictive value of urine pregnancy test CHECK TOP taking as reference transvaginal ultrasound.
  A negative result at transvaginal ultrasound will be defined as the absence of ongoing pregnancy. An ongoing pregnancy is characterized by the presence of gestational sac, yolk sac and/or embryo with cardiac activity. A positive result will be retained only in case of ongoing pregnancy.
  Check Top test will be considered as negative if only one colored line appears in the control window, without any line in the result window. It will be considered as positive if two colored lines are present in the result window, corresponding to a β-HCG level > 1000 IU/ml.

SECONDARY OUTCOMES:
Positive predictive value of urine pregnancy test Check Top | During control visit post drug abortion, after transvaginal ultrasound (at day14 or day21)
  Positive predictive value of urine pregnancy test Check Top compared to transvaginal ultrasound.
Sensibility of urine pregnancy test Check Top | During control visit post drug abortion, after transvaginal ultrasound (at day14 or day21)
  Sensibility of urine pregnancy test Check Top compared to transvaginal ultrasound.
Specificity of urine pregnancy test Check Top | During control visit post drug abortion, after transvaginal ultrasound (at day14 or day21)
  Specificity of urine pregnancy test Check Top compared to transvaginal ultrasound.
Acceptability of urine pregnancy test Check Top by patients. | During control visit post drug abortion, after transvaginal ultrasound (at day14 or day21)
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon, France